CLINICAL TRIAL: NCT01006213
Title: Group Motivational Intervention in Overweight/Obese Patients in Primary Prevention of Cardiovascular Disease in the Primary Healthcare Area (IMOAP)
Brief Title: Group Motivational Intervention in Overweight/Obese Patients
Acronym: IMOAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Jordi Gol i Gurina Foundation, IDIAP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI070087
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Overweight; Obesity
Keywords: Motivational Intervention
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling vs motivational intervention (Experimental)
  Interventions: Behavioral: Motivational intervention

INTERVENTIONS:
Behavioral: Motivational intervention — Two groups will be established in geographically separate areas, one of which will receive the group motivational intervention (intervention group) and the other will receive standard follow-up (control group)

SUMMARY:
Overall mortality, such as that caused by cardiovascular disease, increases as weight increases. In the Framingham Study, it was shown that obesity is a cardiovascular risk factor independent of other risk factors such as type 2 diabetes mellitus, dyslipidemia and smoking.

Objectives:

1. To determine whether a group motivational intervention is more effective than the standard intervention for treatment of overweight and obesity and most importantly to maintain the attained weight loss on a permanent basis.
2. To assess whether this intervention is more effective than reducing cardiovascular risk factors (lipid profile, apo B-100, apo A-1, fibrinogen, C-reactive protein, hypertension, diabetes mellitus) associated with overweight and obesity, and the overall cardiovascular risk in these patients.

Design: Randomized, multicenter, interventional clinical trial in patients with overweight and obesity. Randomized assignment of the intervention by Basic Health Areas (BHAs). Two groups will be established in geographically separate areas, one of which will receive the group motivational intervention (intervention group) and the other will receive standard follow-up (control group). BHAs located in the same building will be assigned the same group (control or intervention) to avoid potential contamination. hypertensive treatment or with a diagnosis of hypertension in their clinical history.

Study Scope: Primary care. The study will be conducted in 24 BHAs of Hospitalet de Llobregat and Barcelona during 26months follow-up period. Haematic analyses will be in the carried out at the reference laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI>25) and obese (BMI>30) patients of both sexes, registered in the medical history (MH) or newly diagnosed.
* Aged between 30 and 70 years
* Agreement to participate in the study

Exclusion Criteria:

* Patients with severe clinical pathology (bedridden, dementia, advanced neoplasia, etc.)
* Patients with secondary obesity (hypothyroidism, Cushing's disease, etc).
* Patients with severe sensorial disorders capable of interfering with the motivational intervention
* Patients with serious psychiatric disorders

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-01 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
If a group of motivational intervention, together with current clinical practice, is more efficient than the latter in the treatment of overweight and obesity | two years

SECONDARY OUTCOMES:
Observe whether this intervention is more effective for reducing cardiovascular risk factors (lipid profile, apo B-100, apo A-1, fibrinogen, reactive protein C, hypertension, diabetes mellitus) | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Abs Florida Sur, L'Hospitalet de Llobregat, BARCELONA, Spain

REFERENCES:
- [Derived] Rodriguez-Cristobal JJ, Alonso-Villaverde C, Panisello JM, Trave-Mercade P, Rodriguez-Cortes F, Marsal JR, Pena E. Effectiveness of a motivational intervention on overweight/obese patients in the primary healthcare: a cluster randomized trial. BMC Fam Pract. 2017 Jun 20;18(1):74. doi: 10.1186/s12875-017-0644-y. PMID 28633627
- [Derived] Rodriguez Cristobal JJ, Alonso-Villaverde Grote C, Trave Mercade P, Perez Santos JM, Pena Sendra E, Munoz Lloret A, Fernandez Perez C, Bleda Fernandez D; EFAP group. Randomised clinical trial of an intensive intervention in the primary care setting of patients with high plasma fibrinogen in the primary prevention of cardiovascular disease. BMC Res Notes. 2012 Mar 1;5:126. doi: 10.1186/1756-0500-5-126. PMID 22381072
- [Derived] Rodriguez Cristobal JJ, Panisello Royo JM, Alonso-Villaverde Grote C, Perez Santos JM, Munoz Lloret A, Rodriguez Cortes F, Trave Mercade P, Benavides Marquez F, Marti de la Morena P, Gonzalez Burgillos MJ, Delclos Baulies M, Bleda Fernandez D, Quillama Torres E; IMOAP Group. Group motivational intervention in overweight/obese patients in primary prevention of cardiovascular disease in the primary healthcare area. BMC Fam Pract. 2010 Mar 18;11:23. doi: 10.1186/1471-2296-11-23. PMID 20298557